CLINICAL TRIAL: NCT03824093
Title: High and Low Resource Interventions to Promote HPV Vaccines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of Kansas Medical Center (Other); Midwest Cancer Alliance (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ChildrensMHC
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Human Papilloma Virus; Tdap - Tetanus, Diphtheria and Acellular Pertussis Vaccination; Meningitis, Meningococcal; Communication; Satisfaction
Keywords: Adolescent Vaccines
MeSH Terms: conditions — Diphtheria; Meningitis, Meningococcal; Communication; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant
Masking Description: Practices will be randomly assigned to the AFIX only or AFIX+ communication training study arms. Both groups will receive identical AFIX consultations, but only practices assigned to the AFIX+ communication training arm will receive brief, provider communication training and commitment poster displays. Once practices have been randomized, parents of adolescent patients will be exposed to one of the interventions based on their practice location. Participants will not be informed of their practice's study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AFIX Only (Active Comparator): Practices enrolled in the AFIX only arm will receive an in-person AFIX consultation that includes assessment of current HPV vaccination rates and feedback on strategies to increase vaccination rates.
  Interventions: Behavioral: AFIX Only
- AFIX+ Provider Communication Training (Active Comparator): Practices enrolled in the AFIX+ Provider Training arm will receive an in-person AFIX consultation along with a brief communication training for providers and poster and brochure displays in clinic waiting and exam rooms.
  Interventions: Behavioral: AFIX+ Provider Communication Training

INTERVENTIONS:
Behavioral: AFIX Only — The intervention will include an in-person AFIX assessment of the practice's adolescent vaccination rates.
  Arms: AFIX Only
Behavioral: AFIX+ Provider Communication Training — The intervention will include an in-person AFIX assessment of the practice's adolescent vaccination rates along with communication training for providers and poster and brochure displays.
  Arms: AFIX+ Provider Communication Training

SUMMARY:
Human Papillomavirus (HPV) is a significant public health issue affecting nearly 14 million people in the United States. HPV can lead to cervical, oropharyngeal, anal, and penile cancers as well as genital warts.The purpose of this study is to test the comparative effectiveness of two interventions, AFIX only vs. AFIX + communication training, to increase Human Papillomavirus (HPV) vaccination rates among adolescent patients in outpatient clinic settings. Providers and staff at four pediatric practices will be randomized to receive an in-person AFIX consultation or an AFIX consultation combined with communication training and commitment poster displays. Provider and parent data will be collected via a tablet computer RedCap survey. Additional practice and provider level HPV vaccination rates will be collected via patient de-identified claims data. The results of this study could contribute to the existing body of literature that suggests provider recommendations and routine vaccination assessments are key to increasing HPV vaccination uptake. This project has the potential to lead to the implementation and dissemination of low resource interventions to increase HPV vaccination rates among children and adolescents.

DETAILED DESCRIPTION:
Significance: Human Papillomavirus (HPV) is the most common sexually transmitted infection in the United States with an estimated 14 million new infections each year. While most HPV infections resolve without any symptoms or signs of infection, some HPV infections can lead to genital warts and cancer. Every year, more than 30,000 people are affected by an HPV-related cancer, including cervical, oropharyngeal, vaginal and anal cancers. Because most adults will become infected with HPV at some point in their lives, the CDC recommends routine vaccination for girls aged 11-26 and boys aged 11-21. While vaccines to prevent HPV infection have been widely available for more than a decade nearly 38% of eligible girls and 50% of eligible boys have not initiated the HPV vaccine series and more than 70% of boys and 50% of girls have not completed the full vaccine series. Rates of HPV vaccination are significantly lower than rates for other adolescent recommended vaccines including, tetanus, diptheria, and acellular pertussis (Tdap), and meningococcal conjugate (MenACWY), which range from 81 to 86 percent. There are many factors that contribute to less than optimal HPV vaccination rates but chief among them is lack of a strong provider recommendation to initiate and complete the HPV vaccine series.

Innovation: This study will be the first randomized controlled trial comparing the effectiveness of an AFIX intervention vs. an AFIX intervention combined with a provider "nudge" that includes a brief communication skills training and commitment messaging displays to increase HPV vaccination rates in pediatric outpatient settings.

Approach: 200 eligible parents (or caregivers) of adolescents between the ages of 11 and 18 will be enrolled and exposed to one of the interventions based on their clinic location. Parents will be recruited from the Children's Mercy Hospital Primary Care Clinic (CMH PCC) and Cradle Thru College Care Pediatrics in Kansas City, MO, Preferred Pediatrics in Lee's Summit, MO, and Cass County Pediatrics in Belton,MO. Practices will be randomized to receive either an in-person AFIX assessment or an in-person AFIX assessment combined with a brief, provider communication training and adolescent vaccine commitment poster displays. The primary outcome of this study is HPV vaccination rates. A secondary outcome is parent ratings of satisfaction with their child's visit with the health care provider. Data will be collected via a tablet computer administered RedCap survey in the exam room immediately following the child's visit.

Public Health Impact: This study could have a significant public health impact and contribute to meeting the Healthy People 2020 goals to reduce vaccine preventable infections by increasing vaccination rates in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian of a child 11-18 years of age or a pediatric health care provider
* Parent or legal guardian of a child being seen for a well-child visit
* Ability to provide informed consent

Exclusion Criteria:

* Prior participation in the study
* Unable to read or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

PRIMARY OUTCOMES:
HPV vaccination rates | 18 months
  Practice and provider level HPV vaccination rates will be collected from patient de-identified claims data.

SECONDARY OUTCOMES:
Parent Satisfaction | 18 months
  Parent satisfaction with visit will be collected using validated measures on tablet computers

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospital Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
We will create a clean, de-identified copy of our final dataset that will be available to other researcher groups, upon request, within 9 months of the end of the study period. Prior to data sharing, we will remove all identifying information. We will make data and associated documentation available to users under a data-sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available 9 months after the conclusion of the study upon request and completion of a data sharing agreement.